CLINICAL TRIAL: NCT03612557
Title: A Phase 1, Open-label Study To Investigate The Pharmacokinetics And Safety Of A Single Intramuscular Injection Of Benzathine Benzylpenicillin In Japanese Healthy Subjects
Brief Title: A Study of Benzathine Benzylpenicillin Intramuscular Injection in Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B8441001
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Benzathine benzylpenicillin; penicillin G benzathine
MeSH Terms: interventions — Penicillin G Benzathine; Penicillin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- active treatment arm (Experimental): penicillin G benzathine treatment
  Interventions: Drug: penicillin G benzathine

INTERVENTIONS:
Drug: penicillin G benzathine — 2.4 million units (IM) of benzathine benzylpenicillin
  Other Names: penicillin G; benzathine benzylpenicillin

SUMMARY:
This will be an open label study to investigate the pharmacokinetics (PK) and safety of a single intramuscular injection of penicillin G benzathine in Japanese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects (of childbearing or nonchildbearing potential) and/or male subjects
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg and <100 kg.

Exclusion Criteria:

• Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (history of penicillin hypersensitivity and/or a history of sensitivity to allergens).

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration for penicillin G (Cmax) | 0, 3, 6, 12, 24, 36, 48, 144, 312, 480, and 648 hours post dose
Time to Cmax (Tmax) | 0, 3, 6, 12, 24, 36, 48, 144, 312, 480, and 648 hours post dose
Area under the plasma concentration time curve from time zero to the time of the last measurable concentration (AUClast) | 0, 3, 6, 12, 24, 36, 48, 144, 312, 480, and 648 hours post dose
Area under the plasma concentration time curve from time zero extrapolated to infinite time (as data permit)(AUCinf) | 0, 3, 6, 12, 24, 36, 48, 144, 312, 480, and 648 hours post dose
Apparent clearance (as data permit) (CL/F) | 0, 3, 6, 12, 24, 36, 48, 144, 312, 480, and 648 hours post dose
Apparent volume of distribution (as data permit) (Vz/F) | 0, 3, 6, 12, 24, 36, 48, 144, 312, 480, and 648 hours post dose
Terminal half life (as data permit) (t1/2) | 0, 3, 6, 12, 24, 36, 48, 144, 312, 480, and 648 hours post dose

SECONDARY OUTCOMES:
Number of Subjects experiencing an Adverse Event | Screening up to 28 days after last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- P-one Clinic, Keikokai Medical Corporation, Hachioji-shi, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B8441001&StudyName=A+Phase+1%2C+Open-label+Study+To+Investigate+The+Pharmacokinetics+And+Safety+Of+A+Single+Intramuscular+Injection+Of+2%2C400%2C000+Units+Penicillin+G+Benzathine+In+Japanese+Healthy+Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B8441001&StudyName=A+Phase+1%2C+Open-label+Study+To+Investigate+The+Pharmacokinetics+And+Safety+Of+A+Single+Intramuscular+Injection+Of+Benzathine+Benzylpenicillin+In+Japanese+Healthy+Subjects